CLINICAL TRIAL: NCT06291285
Title: A Study to Investigate the Pharmacokinetics and Pharmacodynamics of a Single Oral Dose of Decitabine and Tetrahydrouridine (NDec) When Administered Either as a Modified Release Formulation or an Immediate Release Formulation in Healthy Participants
Brief Title: A Study to Test How Either a Capsule or a Tablet With NDec (Decitabine and Tetrahydrouridine) Works in the Body of Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NN7533-7587; U1111-1285-7491 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Formulation A followed by Formulation B (Experimental): Participants will receive a single oral dose of decitabine and tetrahydrouridine (THU) immediate release tablets (Formulation A) on Day 1 of treatment period 1 followed by a single oral dose of decitabine and THU delayed release capsules (Formulation B) on Day 1 of treatment period 2. A washout period of 7- 21 days will be maintained between the two treatment periods.
  Interventions: Drug: Decitabine-THU
- Formulation B followed by Formulation A (Experimental): Participants will receive a single oral dose of decitabine and THU delayed release capsules (Formulation B) on Day 1 of treatment period 1 followed by a single oral dose of decitabine and THU immediate release tablets (Formulation A) on Day 1 of treatment period 2. A washout period of 7- 21 days will be maintained between the two treatment periods.
  Interventions: Drug: Decitabine-THU

INTERVENTIONS:
Drug: Decitabine-THU — Orally administered immediate release tablets.
  Other Names: NDec
Drug: Decitabine-THU — Orally administered delayed release capsules.
  Other Names: NDec

SUMMARY:
This study will look at two different oral formulations and compare them. The medicine in the study is called NDec and it is a combination of two medicines (decitabine and tetrahydrouridine). Both medicines are new for the treatment of sickle cell disease, a rare blood disease. The purpose of the study is to compare the absorption of two different NDec versions (a tablet and a capsule). Participant will either get first the tablet and then the capsule, or the other way around. The order in which participant get them is decided by chance. The study will last for about 12 to 45 days depending on the wash-out period between the two stays in the clinic and from recruitment to the first study day.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female.
* Age 18 64 years (both inclusive) at the time of signing the informed consent.
* Body weight between 60.0 and 100.0 kilogram (kg) (both inclusive) at screening.
* Body mass index between 18.5-29.9 kilograms per square meter (kg/m^2) (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Platelet count greater than (>) 400*10^9/ Liter (L) at visit 1
* Absolute neutrophil count less than or equal to (≤) 1.5*10^9/L at visit 1
* Female who is:

  1. pregnant, breast-feeding or intends to become pregnant during the trial or within 6 months after the last dose of trial product or
  2. of childbearing potential and not using highly effective contraceptive method and whose male partner is not using effective contraception, from screening until 6 months after the last dose of trial product
* Male of reproductive age with female partner of childbearing potential who does not agree to use condoms and whose female partner of childbearing potential is not using a highly effective contraceptive measure (or adequate contraceptive measure as required by local regulation or practice) from signing the informed consent form (ICF) until 6 months after the last dose.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
AUC0-inf,DEC,SD: Area under the plasma decitabine concentration-time curve after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in hours*nanogram per milliliter (h*ng/mL).

SECONDARY OUTCOMES:
AUC0-inf,THU,SD: Area under the plasma tetrahydrouridine concentration-time curve after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in h*ng/mL.
Cmax,DEC,SD: Maximum plasma concentration of decitabine after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in nanogram per milliliter (ng/mL).
Cmax,THU,SD: Maximum plasma concentration of tetrahydrouridine after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in ng/mL.
t½,DEC,SD: Terminal half-life for decitabine after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in hours.
t½,THU,SD: Terminal half-life for tetrahydrouridine after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in hours.
tmax,DEC,SD: Time to maximum observed plasma decitabine concentration after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in hours.
tmax,THU,SD:: Time to maximum observed plasma tetrahydrouridine concentration after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in hours.
Maximum change from pre dose in dNA methyltransferase 1 (DNMT1) protein expression after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in mean fluorescence intensity (MFI).
Maximum change from pre dose in cytidine deaminase (CDA) activity after a single dose | Predose (Day 1) up to 48 hours post dose (Day 3)
  Measured in micromoles per liter per minute (µmol/L/min).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- ICON-Salt Lake City, Salt Lake City, Utah, United States
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com